CLINICAL TRIAL: NCT00072163
Title: A Phase II Study Of Temozolomide And Thalidomide In Patients With Metastatic Melanoma In The Brain
Brief Title: Temozolomide and Thalidomide in Treating Patients With Brain Metastases Secondary to Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02560; CALGB-500102; U10CA031946 (NIH); CDR0000335518 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma; Tumors Metastatic to Brain
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — Temozolomide; Thalidomide

ARMS (1):
- Treatment (temozolomide, thalidomide) (Experimental): Patients receive oral temozolomide once daily on days 1-42 and oral thalidomide once daily on days 1-56. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity. Patients achieving CR receive 2 additional courses of therapy beyond CR.
  Interventions: Drug: temozolomide; Drug: thalidomide

INTERVENTIONS:
Drug: temozolomide — Given orally
  Other Names: SCH 52365; Temodal; Temodar; TMZ
Drug: thalidomide — Given orally
  Other Names: Kevadon; Synovir; THAL; Thalomid

SUMMARY:
This phase II trial is studying how well giving temozolomide together with thalidomide works in treating patients with brain metastases secondary to melanoma. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop tumor cells from dividing so they stop growing or die. Thalidomide may stop the growth of cancer by stopping blood flow to the tumor. Combining temozolomide with thalidomide may kill more tumor cells

DETAILED DESCRIPTION:
OBJECTIVES: Primary I. Determine the objective response rate in patients with brain metastases secondary to melanoma treated with temozolomide and thalidomide.

Secondary I. Determine the toxic effects of and tolerance to this regimen in these patients.

II. Determine the objective response rate in extracranial metastases of patients treated with this regimen.

III. Determine the time to first disease progression (intra- or extracranial) in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive oral temozolomide once daily on days 1-42 and oral thalidomide once daily on days 1-56. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity. Patients achieving complete response (CR) receive 2 additional courses of therapy beyond CR.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually for up to 2 years.

PROJECTED ACCRUAL: A total of 21-50 patients will be accrued for this study within 1.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic melanoma
* Clinical evidence of brain metastases

  * At least 1 unidimensionally measurable brain lesion at least 2.0 cm by conventional techniques OR at least 1.0 cm by spiral CT scan or MRI

    * The following lesions are not considered measurable:

      * Bone lesions
      * Leptomeningeal disease
      * Ascites
      * Pleural/pericardial effusion
      * Lymphangitis cutis/pulmonis
      * Abdominal masses that are not confirmed and followed by imaging techniques
      * Cystic lesions
      * Lesions situated in a previously irradiated area, unless new growth is documented
* Performance status - CTC 0-1
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* AST and ALT no greater than 2.5 times upper limit of normal (ULN)
* Lactic dehydrogenase no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* Creatinine no greater than 2 mg/dL
* No history of active angina
* No history of significant ventricular arrhythmia
* No history of deep vein thrombosis
* No myocardial infarction within the past 6 months
* No acute abnormality by EKG
* No uncontrolled arrhythmia
* No history of pulmonary embolism
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 1 highly-effective and 1 additional method of contraception for 28 days before, during, and for 4 weeks after study participation
* No known HIV disease
* Thyroid-stimulating hormone normal
* Serum anticonvulsant levels normal (for patients on anticonvulsants)
* No frequent vomiting and/or any other medical condition (e.g., partial bowel obstruction) that would preclude oral medication intake
* No preexisting neuropathy greater than grade 1
* No uncontrolled seizures
* No other concurrent medical condition that would preclude study participation
* At least 4 weeks since prior cytokines

  * Biologic agents used as adjuvants, vaccines, and cellular therapies do not require a 4-week washout period
* No concurrent prophylactic filgrastim (G-CSF) or sargramostim (GM-CSF)
* No more than 1 prior chemotherapy regimen
* No prior chemotherapy for brain metastases
* No prior continuous daily temozolomide
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No other concurrent chemotherapy
* No concurrent hormonal therapy except steroids and hormones administered for non-disease-related conditions (e.g., insulin for diabetes) or for control of intracranial edema from brain metastases
* See Disease Characteristics
* Prior whole brain radiotherapy (WBRT) allowed provided patient has progressive disease in a measurable CNS lesion
* Prior stereotactic radiotherapy allowed provided patient has progressive disease in a measurable CNS lesion
* At least 4 weeks since prior WBRT
* At least 3 weeks since prior stereotactic radiosurgery
* No concurrent radiotherapy
* At least 3 weeks since prior surgical resection
* No concurrent warfarin or heparin products or their derivatives
* No concurrent antiplatelet therapy (e.g., daily aspirin, ibuprofen, or clopidogrel bisulfate)
* No concurrent bisphosphonates (e.g., zoledronate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-10; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Response rate (defined as complete or partial) | Up to 5 years
  90% confidence intervals will be used.

SECONDARY OUTCOMES:
Time to first progression | Up to 5 years
  Kaplan-Meier method will be used.
Overall survival | Up to 5 years
  Kaplan-Meier method will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Krown, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States